CLINICAL TRIAL: NCT04852133
Title: Feasibility and Reliability of Ultrasound Assessment of Muscle Architecture in Acute Burns.
Brief Title: Feasibility and Reliability of Ultrasound in Acute Burns.
Status: Completed | Type: Observational
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Principal Investigator, Ulrike Van Daele, Full Professor, Universiteit Antwerpen
Other Study IDs: 11B8619N[US]
Record Dates: First submitted 2021-04-15; First posted 2021-04-21 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Burns
Keywords: Burns; Ultrasound; Muscle wasting; Muscular Atrophy; Reliability; Feasibility
MeSH Terms: conditions — Burns; Muscular Atrophy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Burn subjects: exposure to burn injury
  Interventions: Other: Burn subjects
- Non-burned control: no exposure to burn injury

INTERVENTIONS:
Other: Burn subjects — see eligibility criteria
  Groups: Burn subjects

SUMMARY:
This trial investigates the feasibility and reliability of different ultrasound protocols to determine quadriceps muscle architecture in acutely admitted burn patients. The results of this trial will provide more clarity as to whether ultrasound can be used as a bedside tool to monitor muscle wasting.

DETAILED DESCRIPTION:
BACKGROUND Despite the ubiquity of muscle wasting following burns, practical and accurate tools to measure the degree of muscle wasting are lacking in burn care. Ultrasound has been used for this purpose in the critically-ill population and has shown to be valid and reliable. Whether this can be extrapolated to the burn population, however, remains unclear. Open wounds, fluid status, and uncertainty regarding which protocol to use are amongst factors that complicate the use of ultrasound during the acute phase of burns.

AIM This study examines the reliability and feasibility of ultrasound measures in the acute burn setting comparing different techniques and locations of application.

METHODS Burned adults were assessed at admission in two Belgian burn centers by two trained assessors using B-mode ultrasound with a linear transducer. Ultrasound-derived variables included quadriceps muscle layer thickness (QMLT) and rectus femoris cross-sectional area (RF-CSA) on both thighs. Both maximum and minimum compression techniques were used for QMLT, while RF-CSA was determined by minimum compression only. QMLT was measured at a proximal and distal location on the thigh, and RF-CSA was measured at the most proximal location possible where the entire muscle belly still remained visible.

ELIGIBILITY:
Burn subjects:

Inclusion Criteria:

* ≥10 - ≤80 %TBSA
* Burn depth: 2nd deep / 3rd degree

Exclusion Criteria:

* Electrical burn (except flash burns)
* Associated injury: fracture lower limb
* Diabetes Mellitus type 1
* Central / peripheral neurological/neuromuscular disorders (interfering with exercise)
* Cognitive / psychological disorders (interfering with cooperation)
* Cardiopulmonary disease (interfering with exercise safety)
* Pregnancy
* Palliative care

Healthy subjects:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Burn subjects will be recruited from two specialised burn services in Belgium on a consecutive sampling basis during recruitment of a larger trial investigating the effects of exercise in the acute phase of burns [NCT04511104].
  Healthy subjects will be recruited by convenience sampling at the M2Run Metabolic Research Unit of the Department of Rehabilitation Sciences and Physiotherapy at the University of Antwerp.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-04-06 (Actual)

PRIMARY OUTCOMES:
Reliability | <72 hours of admission
  Interrater reliability of QMLT and RF-CSA assessed by intraclass correlation

SECONDARY OUTCOMES:
Feasibility of measurements | <72 hours of admission
  Feasibility of different techniques and locations of measurements, assessed by number of realised vs attempted measurements

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Van Daele, PhD, Principal Investigator — University of Antwerp, Faculty of Medicine and Health Sciences
Locations (2):
- Belgium (2):
  - Ziekenhuis Netwerk Antwerpen Stuivenberg, Antwerp
  - Militaire Hospitaal Koningin Astrid, Neder-Over-Heembeek, Brussels

IPD SHARING:
Plan to Share IPD: No
Datasets will be made available upon request.